CLINICAL TRIAL: NCT01231230
Title: Interactive Acute Smooth Muscle Effects of Salmeterol and Fluticasone in the Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 20060346
Record Dates: First submitted 2010-10-25; First posted 2010-11-01 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
Keywords: asthma, corticosteroids, bronchodilator, airway blood flow
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Sugars; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- fluticasone/salmeterol (Experimental): participants were treated fluticasone/salmeterol,
  Interventions: Drug: fluticasone/salmeterol
- salmeterol (Experimental): participants were treated with salmeterol
  Interventions: Drug: Salmeterol
- fluticasone (Experimental): participants were treated with fluticasone
  Interventions: Drug: fluticasone
- placebo inhalation (Placebo Comparator): participants were treated with placebo
  Interventions: Drug: placebo inhalation

INTERVENTIONS:
Drug: fluticasone — 220- mcg once
  Other Names: flovent
  Arms: fluticasone
Drug: placebo inhalation — placebo inhalation once
  Other Names: sugar pill
  Arms: placebo inhalation
Drug: Salmeterol — 50 mcg salmeterol once
  Other Names: serevent
  Arms: salmeterol
Drug: fluticasone/salmeterol — inhalation of 250 mcg of fluticasone combined with 50 mcg of salmeterol
  Other Names: advair
  Arms: fluticasone/salmeterol

SUMMARY:
The addition of an inhaled long-acting beta-adrenergic agonist to an inhaled glucocorticosteroid improves disease control in persistent asthma. This observation has supported the use of long-acting beta-adrenergic agonist/glucocorticosteroid combination preparations for the management of asthma. Currently, salmeterol/fluticasone and formoterol/budesonide are available for clinical use. The long-term beneficial clinical effects of the two drug classes seem to be synergistic, and several mechanisms of glucocorticoid-beta-adrenergic agonist interactions involving gene transcription have been invoked to explain this phenomenon.This study, wish to address the question whether glucocorticoids can acutely potentiate the bronchodilator response to a long-acting beta-adrenergic agonist.We expect that in patients with asthma, the short-term bronchodilator effect of salmeterol is enhanced by the addition of fluticasone, which by itself has no short-term bronchodilator effect. To test this premise, we will assess the respective short-term effects of salmeterol (50 µg), fluticasone (250 µg), salmeterol/fluticasone (50/250 µg), and placebo/placebo on spirometric parameters. Airway Blood flow will also be measured to ensure that vasoconstriction does not occur.

DETAILED DESCRIPTION:
Fourteen lifetime nonsmokers with a physician diagnosis of asthma will be recruited for the study. All subjects will be allowed to use short-acting beta-adrenergic agonists as rescue medication.

Inclusion criteria:

1. Males and females, 18 to 65 years of age.
2. FEV1 60-85% of predicted on the screening day.

Exclusion criteria:

1. Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women.
2. Cardiovascular disease and/or use of cardiovascular medications

2. Subjects with known beta-adrenergic agonist or glucocorticosteroid intolerance 4. Acute respiratory infection within four weeks prior to the study 5. Use, within two weeks prior to the study, of any anti-asthma medication not mentioned above

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 to 65 years of age.
2. FEV1 60-85% of predicted on the screening day. -

Exclusion Criteria:

1. Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women. 2. Cardiovascular disease and/or use of cardiovascular medications 3. Subjects with known beta-adrenergic agonist or glucocorticosteroid intolerance 4. Acute respiratory infection within four weeks prior to the study 5. Use, within two weeks prior to the study, of any anti-asthma medication not mentioned above

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendes ES, Rebolledo P, Wanner A. Acute effects of salmeterol and fluticasone propionate alone and in combination on airway blood flow in patients with asthma. Chest. 2012 May;141(5):1184-1189. doi: 10.1378/chest.11-0685. Epub 2011 Oct 6. PMID 21980058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from our Asthma Database. Subjects with asthma who are in our database have previously agreed to serve as potential subjects in future studies. These subjects have signed an informed consent (approved by UM IRB) to be included in this database.
Groups:
- All Study Groups: inhalation of 250 mcg of fluticasone
  fluticasone: 220- mcg once
Period: Overall Study
Arm/Group | All Study Groups
Started | 14
Fluticasone | 14
Salmeterol | 14
Fluticasone/Salmeterol | 14
Placebo | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fourteen lifetime nonsmokers with a physician diagnosis of asthma were recruited for the study. All but one of the subjects were using an ICS/LABA combination preparation regularly, and all used a short-acting b2-adrenergic agonist as rescue medication. All subjects had to have a prebronchodilator FEV1 of 60% to 85% predicted .
Groups:
- All Study Participants: participant received in random order one of the four treatments ( fluticasone, salmeterol, fluticasone+salmeterol or placebo)
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Airway blood flow (Qaw) [Mean (Standard Deviation); unit: µl.min-1.ml-1] — Qaw was measured with a previously validated soluble inert gas uptake method. It is based on quantifying the disappearance of the soluble gas dimethylether (DME) from the anatomical dead space. The method involves the inhalation of a gas mixture containing 10 % DME and 90% nitrogen from 500 ml below the total lung capacity position to total lung capacity, followed by a breathhold (5 or 15 sec) and subsequent exhalation while the instantaneous concentrations of DME and nitrogen are recorded.
  µl.min-1.ml-1 | 54.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in Airway Blood Flow (Qaw)
Time Frame: maximum change in Qaw within 240 minutes post drug inhalation
Measure: Mean (Standard Error); unit: change from baseline ( µl/min/ml)
Groups:
- Fluticasone: inhalation of 250 mcg of fluticasone
  fluticasone: 220- mcg once
- Placebo: inhalation of placebo diskus
  placebo inhalation: placebo inhalation once
- Salmeterol: inhalation of salmeterol 50 mcg once
  Salmeterol: 50 mcg salmeterol once
  Salmeterol: 50 mcg once
- Fluticasone/Salmeterol: inhalation of fluticasone 250mcg combined with salmeterol 50 mcg
  fluticasone/salmeterol: inhalation of 250 mcg of fluticasone combined with 50 mcg of salmeterol
Arm/Group | Fluticasone | Placebo | Salmeterol | Fluticasone/Salmeterol
Number analyzed (Participants) | 14 | 14 | 14 | 14
change from baseline ( µl/min/ml) | -11.0 (2.9) | 14.1 (1.9) | 23.9 (3.6) | 25.5 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone/Salmeterol; mean difference from baseline relative to placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 15
Statistical Analysis 2: Comparison: Placebo vs Salmeterol; mean difference from baseline relative to placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Fluticasone vs Placebo; mean difference from baseline relative to placebo; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Fluticasone | Placebo | Salmeterol | Fluticasone/Salmeterol
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes